CLINICAL TRIAL: NCT06461598
Title: Development and Validation of the ChemoResist Signature Precisely Predictive of Chemotherapy Sensitivity in Resected Pancreatic Ductal Adenocarcinoma
Brief Title: Signature for Precise Chemosensitivity Prediction in PDAC
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, lei huang, PI, Ruijin Hospital
Other Study IDs: ChemoResist-01
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort
  Interventions: Drug: Chemotherapy
- Validation cohort
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — All adjuvant chemotherapy for nonmetastatic PDAC was gemcitabine-based (Cycle >= 1).

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is largely heterogeneous. We sought to develop and validate a signature to precisely predict chemotherapy sensitivity in PDAC. Genetic events of the four most commonly mutated genes in PDAC and expressions of 12 PI3K/AKT/mTOR pathway markers were examined in consecutive patients with PDAC. A 9-feature signature for prediction of chemotherapy benefits was constructed using the LASSO Cox regression model, and validated in two independent cohorts.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status score of 0-1 before resection
* complete clinicopathologic and follow-up data
* availability of formalin-fixed paraffin-embedded (FFPE) specimens of resected primary tumor and hematoxylin and eosin slides with invasive tumor components

Exclusion Criteria:

* any previous history of cancer
* any anticancer therapy prior to resection or adjuvant radiotherapy
* metastatic cases
* major postsurgical complications with Clavien-Dindo Grade ≥2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with incident, primary, microscopically-confirmed nonmetastatic PDAC who underwent resection were initially enrolled.
Sampling Method: Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3-year
  Time between resection and death of any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No